CLINICAL TRIAL: NCT04407663
Title: Outpatient Clinic in Obesity Care During COVID-19 Outbreak: Physically Far, Virtually Near. Brief Correspondence on a Single Center Experience. Cohort Study
Brief Title: Outpatient Clinic in Obesity Care During COVID-19 Outbreak: Physically Far, Virtually Near
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: Telemedicine
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Bariatric Surgery Candidate; Patient Underwent Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Patient: Inclusion criteria were as follows: obese adults (> 18 years of age, BMI> 40 or > 35 with comorbidities) older than 18 years; patients undergoing bariatric surgery within 6 months; patients who required clinical and instrumental control; presence of a caregiver in case of subject with cognitive impairment; patients with a history of bariatric surgery who requested a first outpatients access or established patients who requested an outpatients' visit for an emerging problem.
  Interventions: Other: Telemedicine to remote outpatient visit in bariatric patient

INTERVENTIONS:
Other: Telemedicine to remote outpatient visit in bariatric patient — Patients that referred for the first time to our bariatric center were investigated for anthropometric, psychological and instrumental data in order to evaluate the eligibility for a future bariatric procedure. In established patients, eligibility for tele-consultation was evaluated by three experienced physicians, consulting the stored patients' data. All included patients provided oral informed consent. Patients approached the virtual visit with their personal smart devices, desktop or laptop computer. Medical counselling was performed using a desktop or laptop computer from the Hospital or home in a smart working modality. The video call was carried out using Skype platform by Microsoft®; any document drawn up by the physician was saved as pdf using the Cute Professional™ PDF software, that allows to add passwords and set security options to protect the patients' data.

SUMMARY:
Bariatric patients represent a peculiar and frail subset of subjects, constantly increasing. During the novel coronavirus disease outbreak, for the lockdown of any non-urgent and non-oncological activity, the access to healthcare services was severely limited, according to the International Federation for the Surgery of Obesity and Metabolic Disorders.

DETAILED DESCRIPTION:
The constant and strict follow-up is mandatory in this special subset of patients. Therefore, starting from the telemedicine experience in different medical fields, in our bariatric surgery division we designed and started a dedicated project to follow-up obese patients using remote counselling.

ELIGIBILITY:
Inclusion criteria:

* obese adults (> 18 years of age, BMI> 40 or > 35 with comorbidities) older than 18 years
* patients undergoing bariatric surgery within 6 months
* patients who required clinical and instrumental control
* presence of a caregiver in case of subject with cognitive impairment; patients with a history of bariatric surgery who requested a first outpatients access or established patients who requested an outpatients' visit for an emerging problem.

Exclusion criteria:

* virtual visit decline
* the internet or smart devices unavailability
* need for physical examination or radiological investigations established during a preliminary contact by phone.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 138/175 patients (78.8%) were eligible for telemedicine (66 established patients, 25 undergoing surgery within 30 days and 47 for the first time referred to our center).
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility of telemedicine in outpatient visit in bariatric patients | 2 months
  Telemedicine to follow-up and identify sing or symptom of alarm in patient undergoing bariatric surgery or in established bariatric patients during COVID-19 outbreak

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided